CLINICAL TRIAL: NCT07131891
Title: The Effects of Electronic Cigarette and Traditional Cigarette Consumption Habits on Sleep Quality, Fatigue, Mental Health, and Quality of Life
Brief Title: The Effects of Electronic Cigarette and Traditional Cigarette
Status: Completed | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, Seval Yilmaz, Principal Investigator, Atılım University
Other Study IDs: 6040102411- Cigarette
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Cigarette Addiction
Keywords: electronic cigarette; traditional ciagrette; Sleep Quality; Fatigue; Mental Health
MeSH Terms: conditions — Vaping; Sleep Initiation and Maintenance Disorders; Fatigue; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Electronic cigarette: Electronic cigarette users
  Interventions: Other: Fatigue Severity Scale; Other: Depression, Anxiety and Stress Scale-21; Other: Jenkins Sleep Scale; Other: Epworth Sleepiness Scale; Other: Short Form-36
- Traditional cigarette: Traditional cigarette users
  Interventions: Other: Fatigue Severity Scale; Other: Depression, Anxiety and Stress Scale-21; Other: Jenkins Sleep Scale; Other: Epworth Sleepiness Scale; Other: Short Form-36
- Dual: Both electronic and traditional cigarette users
  Interventions: Other: Fatigue Severity Scale; Other: Depression, Anxiety and Stress Scale-21; Other: Jenkins Sleep Scale; Other: Epworth Sleepiness Scale; Other: Short Form-36
- Control: Those who do not use any tobacco products, whether electronic or traditional
  Interventions: Other: Fatigue Severity Scale; Other: Depression, Anxiety and Stress Scale-21; Other: Jenkins Sleep Scale; Other: Epworth Sleepiness Scale; Other: Short Form-36

INTERVENTIONS:
Other: Fatigue Severity Scale — Individuals' fatigue severity will be assessed using the Fatigue Severity Scale (FSS). The scale consists of nine questions, and participants are asked about their fatigue level over the past week. Questions are scored from 1 to 7 using a Likert-type scale, where 1 corresponds to "strongly disagree" and 7 to "strongly agree," with higher scores indicating greater agreement. The total score is calculated by taking the arithmetic mean of all items, with the highest possible score being 7. Scores of 4 and above indicate pathological fatigue. The validity and reliability of the FSS in Turkish have been previously established.
Other: Depression, Anxiety and Stress Scale-21 — The 21-item Depression, Anxiety, and Stress Scale (DASS-21) will be administered to assess individuals' levels of depression, anxiety, and stress. The original scale was developed by Lovibond with 42 items. Subsequently, Brown et al. validated a shorter form for the same purpose and created the 21-item DASS-21. The Turkish adaptation of the DASS-21 was conducted by Yılmaz et al. The scale measures three subscales-depression, anxiety, and stress-consisting of seven items each. It is a 4-point Likert-type scale, with 0 indicating "Does not apply to me," 1 "Applies to me somewhat," 2 "Generally applies to me," and 3 "Applies to me completely." All items are scored positively, and each subscale is categorized as normal, mild, moderate, severe, or very severe.
  Other Names: DASS-21
Other: Jenkins Sleep Scale — The Jenkins Sleep Scale consists of four questions that assess sleep problems over a four-week period. Each question is scored from 0 to 5, resulting in a total score ranging from 0 to 20, with higher scores indicating greater sleep disturbances.
Other: Epworth Sleepiness Scale — The Epworth Sleepiness Scale (ESS) was developed to assess daytime sleepiness. It consists of eight items, each scored from 0 to 3, yielding a total score ranging from 0 to 24. Higher scores indicate greater daytime sleepiness. The Turkish version of the scale was validated for reliability and accuracy by İzci et al. in 2008..
Other: Short Form-36 — Quality of life will be assessed using the Turkish version of the Short Form-36 (SF-36). The SF-36 assesses quality of life under eight subscales: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. Scores for each subscale are calculated separately, ranging from 0 to 100, with higher scores indicating better health status. A total score is not calculated.

SUMMARY:
The aim of the study is to investigate and compare the effects of traditional cigarette and e-cigarette consumption habits on sleep quality, fatigue, mental health and quality of life.

DETAILED DESCRIPTION:
E-cigarettes are battery-powered devices that vaporize a solution that may or may not contain nicotine. Carcinogens and other toxins in e-cigarettes can have negative effects on physical health, and their potential negative effects on mental health are also a concern. Adults in the US who experience serious psychological distress are reported to be more likely to use traditional cigarettes (tobacco), e-cigarettes, or both than adults without serious psychological distress. A relationship between traditional cigarette smoking and mental illness, including depression, is well-known. Recent studies have also found that depressive symptoms are associated with e-cigarette use. A study comparing the relationship between different cigarette products and depressive symptoms found that dual use (traditional cigarettes and e-cigarettes) in young adults was associated with higher depressive symptoms than single use.

Another mental health factor associated with smoking is sleep health. Nicotine is thought to be the primary mechanism linking traditional cigarette use to sleep disorders, as acute withdrawal during the night can cause uncomfortable and sleep-disrupting physiological symptoms. This relationship is also observed in e-cigarette users. In a study conducted with university students, e-cigarette users reported poorer sleep health compared to non-smokers.

Smoking and e-cigarette use are also known to affect fatigue and quality of life. Cao et al. evaluated non-smokers, traditional cigarette users, e-cigarette users, and dual users in terms of fatigue and quality of life. They reported that non-smokers had the lowest fatigue and highest quality of life among these four groups, while the e-cigarette user group had less fatigue and higher quality of life than the traditional cigarette user group.

Various studies in the literature compare e-cigarette and traditional cigarette users in terms of fatigue, sleep quality, depression, mental health, and quality of life. However, there are insufficient studies evaluating all parameters and investigating the relationships among these parameters. Therefore, we believe that our study will provide valuable contributions to the literature in this area.

Another mental health factor associated with smoking is sleep health. Nicotine is thought to be the mechanism linking traditional cigarette use to sleep disorders, as acute withdrawal during the night can cause uncomfortable and sleep-disrupting physiological symptoms. This relationship is also seen in e-cigarette users. In a study conducted with university students, e-cigarette users reported poorer sleep health compared to non-smokers. Smoking and e-cigarette use are also known to affect fatigue and quality of life. Cao et al. evaluated non-smokers, traditional cigarette users, e-cigarette users, and both in terms of fatigue and quality of life. They reported that non-smokers had the lowest fatigue and highest quality of life among these four groups. The e-cigarette user group had less fatigue and higher quality of life than the traditional cigarette user group. Various studies in the literature compare e-cigarette and traditional cigarette users in terms of fatigue, sleep quality, depression, mental health, and quality of life. However, there are insufficient studies evaluating all parameters and investigating their relationship with each other. Therefore, we believe our study will contribute to the literature in this area.

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals between the ages of 18-65

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female individuals between the ages of 18-65
Sampling Method: Non-Probability Sample
Enrollment: 533 (Actual)
Dates: Start 2025-03-30 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | From enrollment to the end of the assessment period at 2 hours
  Individuals' fatigue severity will be assessed using the Fatigue Severity Scale (FSS). The scale consists of 9 questions. Participants are questioned about their level of fatigue over the past week. Questions are scored from 1 to 7. The Likert-type scale is used, with 1 point representing "strongly disagree" and 7 points representing "strongly agree," with higher scores indicating greater agreement. A net score is obtained by calculating the arithmetic mean of all questions. The highest possible score is 7. Scores of 4 and above indicate pathological fatigue. The validity and reliability study of the FSS has been conducted in the Turkish language.
Jenkins Sleep Scale | From enrollment to the end of the assessment period at 2 hours
  The Jenkins Sleep Scale consists of four questions that assess sleep problems over a 4-week period. Each question is scored from 0 to 5. The total score ranges from 0 to 20 and indicates increasing sleep disturbance.

SECONDARY OUTCOMES:
Depression, Anxiety, and Stress Scale (DASS 21) | From enrollment to the end of the assessment period at 2 hours
  The 21-item "Depression, Anxiety, and Stress Scale (DASS 21)" will be administered to determine individuals' depression, anxiety, and stress levels. The scale was first developed by Lovibond and Lovibond (12) with 42 items. Subsequently, Brown et al. (13) determined that a shorter form was valid enough to perform the same measurement, and the 21-item "Depression, Anxiety, and Stress Scale (DASS 21)" was created. Yılmaz et al. (14) adapted the DASS 21 into Turkish. The scale, which measures depression, stress, and anxiety subscales and consists of 21 questions with 7 items for each subscale, is a 4-point Likert-type scale (0: Does not apply to me, 1: Applies to me somewhat, 2: Generally applies to me, and 3: Applies to me completely). All items on the scale are scored positively, and each subscale is evaluated by classifying it as normal, mild, moderate, severe, and very severe.
Epworth Sleepiness Scale | From enrollment to the end of the assessment period at 2 hours
  This scale was developed to assess daytime sleepiness. It consists of a total of eight items, with four different response options ranging from 0 to 3 for each item, and the total score ranges from 0 to 24. The higher the total score, the greater the individual's degree of daytime sleepiness. The scale's validity and reliability in Turkish was conducted by İzci et al. in 2008.
Short Form-36 | From enrollment to the end of the assessment period at 2 hours
  Quality of life was assessed using the Turkish version of the Short Form 36 (SF-36) (18). The SF-36 assesses quality of life under eight subscales: physical function, physical role difficulty, pain, general health, vitality, social function, emotional role difficulty, and mental health. Scores for each subscale are calculated separately. Subscale scores range from 0 to 100, with higher scores indicating better health. A total score is not calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Seval Yılmaz, PhD, Principal Investigator — Atılım University
Locations (1):
- Atılım University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No